CLINICAL TRIAL: NCT00776997
Title: LINX Reflux Management System Clinical Study Protocol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Torax Medical Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1802
Record Dates: First submitted 2008-10-20; First posted 2008-10-22 (Estimated); Results first posted 2013-11-13 (Estimated); Last update posted 2018-05-04 (Actual); Status verified 2018-03

CONDITIONS: Gastroesophageal Reflux
Keywords: Gastroesophageal Reflux
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Magnetic Sphincter Augmentation (Other): Single-arm study: all subjects were treated with magnetic sphincter augmentation. A subject's baseline measurements prior to sphincter augmentation were compared to post-sphincter augmentation measurements. Subjects served as their own control.
  Interventions: Device: Magnetic Sphincter Augmentation

INTERVENTIONS:
Device: Magnetic Sphincter Augmentation — The area of the lower esophageal sphincter (LES) is accessed using a standard laparoscopic approach. The tubular esophagus, in the area of the LES, is sized and the appropriately sized sphincter augmentation device is placed circumferentially around the esophagus in the area of the LES. After confirming proper placement, the ends of the device are secured. At this point, the implant procedure is complete, laparoscopic instruments are withdrawn and access points are closed.
  Other Names: LINX Reflux Management System; Magnetic Esophageal Sphincter

SUMMARY:
The purpose of the study is to evaluate the safety and effectiveness of the LINX Reflux Management System in the treatment of Gastroesophageal Reflux Disease (GERD).

DETAILED DESCRIPTION:
At present, the primary alternative for GERD patients with an incomplete symptomatic response to proton-pump inhibitors (PPIs) is laparoscopic Nissen fundoplication. This surgical procedure continues to be the prevalent non-medical treatment option for GERD patients, despite several important limitations. First, it is a very traumatic procedure, requiring portions of the stomach to be dissected and then wrapped around the tubular esophagus, creating permanent anatomic alterations. Secondly, it can create significant side effects, such as gas bloat syndrome, the inability to belch and the inability to vomit.

The intent of the LINX System is to allow a surgeon, using existing laparoscopic techniques and instruments, to augment a weak LES and restore the defective barrier at the gastroesophageal junction (GEJ). This defect of the GEJ is the source of abnormal reflux. The LINX device is an expandable string of individual titanium beads with magnetic cores. The device is laparoscopically placed as a ring around the lower esophageal sphincter. The magnetic attraction of the beads augments the esophageal sphincter's ability to resist gastric pressures that cause reflux. At rest, the LINX device encircles the sphincter with each bead resting against an adjacent bead, to avoid compression of the tubular esophagus. When swallowing, higher pressures are created, allowing the magnetic bond between beads to break, and the LINX implant to expand radially. This serves to preserve swallow and other physiologic functions, such as belching and vomiting, and avoids the side effect of post-prandial bloating. The device can be placed with minimal dissection, preserving anatomy, and is also removable, if necessary. This provides important benefits as it preserves the native anatomy, unlike the Nissen procedure.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be at least 18 years of age and at least the minimum Age of Majority according to applicable State or Country Law and must be less than 75 years of age, with a life expectancy > 3 years
* Subject is a suitable surgical candidate, i.e. is able to undergo general anesthesia and laparoscopic surgery
* Documented typical symptoms of gastroesophageal reflux disease (GERD) for longer than 6 months (regurgitation or heartburn which is defined as a burning epigastic or substernal pain which responds to acid neutralization or suppression)
* Patient requires daily proton pump inhibitor or other anti-reflux drug therapy
* Total Distal Ambulatory Esophageal pH must meet the following criteria: pH< 4 for ≥ 4.5% of the time Note: Subjects shall have discontinued any GERD medications for at least 7 days prior to testing.
* Subjects with symptomatic improvement on proton-pump inhibitor (PPI) therapy demonstrated by a GERD-Health-Related Quality of Life (GERD-HRQL) score of ≤ 10 on proton-pump inhibitors and ≥ 15 off PPIs, or subjects with a ≥ 6 point improvement when comparing their on PPI and off PPI GERD-HRQL score
* GERD symptoms, in absence of PPI therapy (minimum 7 days)
* If the subject is of child bearing potential must have a negative pregnancy test within one week prior to implant and must agree to use effective means of birth control during the course of the study
* Subject is willing and able to cooperate with follow-up examinations
* Subject has been informed of the study procedures and the treatment and has signed an informed consent form

Exclusion Criteria:

* The procedure is an emergency procedure
* Currently being treated with another investigational drug or investigational device
* History of gastroesophageal surgery, anti-reflux procedures, or gastroesophageal/gastric cancer
* Any previous endoscopic anti-reflux intervention for GERD
* Suspected or confirmed esophageal or gastric cancer
* Any size hiatal hernia >3cm as determined by endoscopy
* Distal esophageal motility (average of sensors 3 and 4) is less than 35 mmHg peristaltic amplitude on wet swallows or <70% (propulsive) peristaltic sequences
* Esophagitis - Grade C or D (LA Classification)
* Body Mass Index (BMI)>35
* Symptoms of dysphagia more than once per week within the last 3 months.
* Diagnosed with Scleroderma
* Diagnosed with an esophageal motility disorder such as but not limited to Achalasia, Nutcracker Esophagus, or Diffuse Esophageal Spasm or Hypertensive LES
* Subject has a history of or known esophageal stricture or gross esophageal anatomic abnormalities (Schatzki's ring, obstructive lesions, etc.)
* Subject has esophageal or gastric varices
* Subject has history of or known Barrett's esophagus
* Cannot understand trial requirements or is unable to comply with follow-up schedule
* Pregnant or nursing, or plans to become pregnant during the course of the study
* Medical illness (i.e. congestive heart failure) that may cause the subject to be non-compliant with or able to meet the protocol requirements or is associated with limited life expectancy (i.e. less than 3 years)
* Diagnosed psychiatric disorder (e.g. bipolar, schizophrenia, etc.), subjects that exhibit depression that are on appropriate medication(s) are allowable.
* Suspected or known allergies to titanium, stainless steel, nickel or ferrous materials
* Subject has an electrical implant or metallic, abdominal implants

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2008-11; Primary Completion 2010-12 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (14):
- United States (13):
  - USC Keck School of Medicine, Los Angeles, California
  - University of California - San Diego, San Diego, California
  - Mayo Clinic, Jacksonville, Florida
  - Phoebe Putney Memorial Hospital, Albany, Georgia
  - Abbott Northwestern Hospital/MNGI, Minneapolis, Minnesota
  - Washington University - Division of Gastroenterology, St Louis, Missouri
  - University of Rochester Medical Center, Rochester, New York
  - The Ohio State University Medical Center / Center for Minimally Invasive Surgery, Columbus, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Legacy Health System, Portland, Oregon
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - University of Washington Medical Center, Seattle, Washington
  - Gundersen Lutheran Clinic, La Crosse, Wisconsin
- Academic Medical Center, Amsterdam, Netherlands

REFERENCES:
- [Derived] Ganz RA, Edmundowicz SA, Taiganides PA, Lipham JC, Smith CD, DeVault KR, Horgan S, Jacobsen G, Luketich JD, Smith CC, Schlack-Haerer SC, Kothari SN, Dunst CM, Watson TJ, Peters J, Oelschlager BK, Perry KA, Melvin S, Bemelman WA, Smout AJ, Dunn D. Long-term Outcomes of Patients Receiving a Magnetic Sphincter Augmentation Device for Gastroesophageal Reflux. Clin Gastroenterol Hepatol. 2016 May;14(5):671-7. doi: 10.1016/j.cgh.2015.05.028. Epub 2015 Jun 2. PMID 26044316
- [Derived] Ganz RA, Peters JH, Horgan S, Bemelman WA, Dunst CM, Edmundowicz SA, Lipham JC, Luketich JD, Melvin WS, Oelschlager BK, Schlack-Haerer SC, Smith CD, Smith CC, Dunn D, Taiganides PA. Esophageal sphincter device for gastroesophageal reflux disease. N Engl J Med. 2013 Feb 21;368(8):719-27. doi: 10.1056/NEJMoa1205544. PMID 23425164

RESULTS

PARTICIPANT FLOW:
Groups:
- LINX System: All subjects are treated with the LINX System during a laparoscopic surgical procedure. Subjects serve as their own control. Baseline measurements are compared to post-implant measurements.
Period: Overall Study
Arm/Group | LINX System
Started | 100
Completed | 98 (98 subjects evaluated at 12-months. Endpoint analysis based on all subjects treated (n=100))
Not Completed | 2
Not completed — Adverse Event | 2

BASELINE CHARACTERISTICS:
Arm/Group | LINX System
Number analyzed (Participants) | 100
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 90
  >=65 years | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.4 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48
  Male | 52
Region of Enrollment [Number; unit: participants]
  United States | 96
  Netherlands | 4
Percentage of total monitoring time esophageal pH <4 [Mean (Standard Deviation); unit: Percentage of total monitoring time] — At baseline, all subjects were evaluated with esophageal pH monitoring with GERD medications discontinued for at least 7 days using the BRAVO System
  Percentage of total monitoring time | 11.6 (4.7)
Gastroesophageal Reflux Disease-Health-Related Quality of Life (GERD-HRQL) total score [Mean (Standard Deviation); unit: Total Score] — The GERD-HRQL scale was administered at baseline with GERD medications discontinued for at least seven days. GERD-HRQL scale objectively quantifies symptom severity. The GERD-HRQL scale consists of 10 questions with the following Responses Scale:
  0 = No Symptoms
  1. = Symptoms noticeable, but not bothersome
  2. = Symptoms noticeable and bothersome, but not every day
  3. = Symptoms bothersome every day
  4. = Symptoms affect daily activities
  5. = Symptoms are incapacitating, unable to do daily activities
  The worst possible score is 50 based on a response of "5" to all 10 questions.
  Total Score | 26.6 (6.6)
Use of daily proton-pump inhibitors (PPIs) [Number; unit: participants] — At time of enrollment, all medications used by a subject were documented.
  participants | 100
Years of proton-pump inhibitor use [Mean (Standard Deviation); unit: years] | 6.3 (4.8)

OUTCOME MEASURES:

1. Primary Outcome: Rate of Occurrence for Device and Procedure Related Serious Adverse Events (SAEs).
Description: SAE was defined as any untoward medical occurrence, whether related to the study device or procedure or not, that meets one or more of the following criteria:
  * Results in death
  * Is life-threatening
  * Requires subject hospitalization > 24 hours
  * Requires prolongation of an existing hospitalization
  * Results in persistent or significant disability/incapacity
  * Results in fetal distress, fetal death, or a congenital anomaly or birth defect
  * Requires intervention to prevent permanent impairment or damage.
  Outcome measure reports number of subjects with reported events.
Time Frame: through 24 months
Measure: Number; unit: participants
Arm/Group | LINX System
Number analyzed (Participants) | 100
participants | 6

2. Primary Outcome: Normalization of Esophageal Acid Exposure Time or Reduced Total Acid Exposure Time of at Least 50% Compared to the Subject's Baseline Measurement by Esophageal pH Testing.
Description: The analysis cohort for the primary efficacy analysis was the treated population which includes all implanted subjects and was determined through esophageal pH testing.
Time Frame: 12 Months
Measure: Number; unit: participants
Arm/Group | LINX System
Number analyzed (Participants) | 100
participants | 64 (4.8)

3. Secondary Outcome: At Least a 50% Reduction in Gastroesophageal Reflux Disease-Health-Related Quality of Life (GERD-HRQL) Total Score Compared to Baseline
Time Frame: 12 months
Measure: Number; unit: participants
Arm/Group | LINX System
Number analyzed (Participants) | 100
participants | 92 (5.4)

4. Secondary Outcome: Average Daily Proton-pump Inhibitor (PPI) Dosage Reduced by at Least 50% Compared to Baseline
Time Frame: 12 months
Measure: Number; unit: participants
Arm/Group | LINX System
Number analyzed (Participants) | 100
participants | 93

ADVERSE EVENTS:
Arm/Group | LINX System
Serious Adverse Events (participants affected / at risk) | 6/100
Other Adverse Events (participants affected / at risk) | 76/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LINX System (N=100)
Dysphagia (Gastrointestinal disorders) | 3 (3)
Nausea (Gastrointestinal disorders) | 2 (2)
Odynophagia (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2)
Pain (General disorders) | 1 (1) — unknown causality
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LINX System (N=100)
Dysphagia (Gastrointestinal disorders) | 68 (76)
Pain (General disorders) | 24 (25)
Stomach Bloating (Gastrointestinal disorders) | 14 (15)
Nausea (Gastrointestinal disorders) | 7 (8)
Odynophagia (Gastrointestinal disorders) | 8 (8)
Hiccups (General disorders) | 8 (8)
Inability to belch or vomit (Gastrointestinal disorders) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less